CLINICAL TRIAL: NCT05620004
Title: Safety and Efficacy of Bifidobacterium Therapy in Patients With Advanced Liver Cancer Receiving Immunotherapy: a Randomized Controlled, Single-center Clinical Trial
Brief Title: Safety and Efficacy of Bifidobacterium Therapy in Patients With Advanced Liver Cancer Receiving Immunotherapy
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Chan Xie, associate chief physician, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XC4
Record Dates: First submitted 2022-11-02; First posted 2022-11-17 (Actual); Last update posted 2022-11-17 (Actual); Status verified 2022-11

CONDITIONS: Advanced Hepatocellular Carcinoma
Keywords: Advanced Hepatocellular Carcinoma; Immunotherapy; Bifidobacterium

STUDY DESIGN:
Intervention Model Description: Select patients with advanced hepatocellular carcinoma who have been clinically consulted by MDT ,those patients will be treated with carrilizumab and apatinib mesylate,and divide them into two groups randomly .Collect the stool specimens and clinical data from those who will be treated with oral bifidobacterium or without bifidobacterium during immunotherapy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Bifidobacterium Bifidum Oral Product (Experimental): patients with advanced hepatocellular carcinoma who will be treate with carrilizumab and apatinib mesylate plus Bifidobacterium Bifidum Oral Product daily
  Interventions: Drug: Bifidobacterium Bifidum Oral Product
- without Bifidobacterium Bifidum Oral Product (No Intervention): patients with advanced hepatocellular carcinoma who will be treate with carrilizumab and apatinib mesylate without Bifidobacterium Bifidum Oral Product daily

INTERVENTIONS:
Drug: Bifidobacterium Bifidum Oral Product — experimental group use Bifidobacterium Bifidum Oral Product and control group without Bifidobacterium Bifidum Oral Product
  Other Names: LiveCombinedBifidobacterium,LactobacillusandStreptococcusthermophilusTablets,Oral
  Arms: Bifidobacterium Bifidum Oral Product

SUMMARY:
This study plans to observe the changes of liver cancer and immune cell subsets by replicating the high abundance intestinal flora and liver cancer mouse model, reveal the relationship and mechanism of intestinal flora in the immunotherapy of liver cancer, and study the impact on prognosis by regulating the positive correlation of lactic acid bacteria and bifidobacteria of rumen coccus in patients with advanced liver cancer receiving immunotherapy

DETAILED DESCRIPTION:
Select patients with advanced hepatocellular carcinoma who have been clinically consulted by MDT,those patients will be treated with carrilizumab and apatinib mesylate, and divide them into two groups randomly .Collect the stool specimens and clinical data from those who will be treated with oral bifidobacterium or without bifidobacterium during immunotherapy.; Use 16S sequencing to detect the changes in the composition ratio of intestinal flora and the level of galactose acid, judge the response to clinical treatment and establish the relationship curve with clinical treatment efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with HCC diagnosed by pathological histology or cytology or clinically confirmed.
2. Expected survival ≥ 12 weeks.
3. No systemic systemic antitumor therapy against hepatocellular carcinoma prior to the first dose.
4. Child-Pugh liver function rating: Grade A or B (≤7 points).
5. Stage IIIa: regardless of tumor status, with vascular invasion, no extrahepatic metastasis; liver function grade Child-Pugh A/B; PS 0~2, IIIb: regardless of tumor status, regardless of vascular invasion, with extrahepatic metastasis; liver function grade Child-Pugh A/B; PS 0~2. Not Stage B not suitable for radical surgery and/or local treatment.
6. ECOG physical status score ≤2.
7. At least one measurable lesion according to RECIST v1.1 (measurable lesion spiral CT tracing length ≥ 10 mm or enlarged lymph node short diameter ≥ 15 mm)
8. Routine blood tests: (no blood transfusion, G-CSF medication correction within 14 days prior to screening)
9. Laboratory test values within 7 days prior to enrollment meet the following requirements (no blood components, cell growth factors, albumin, or other corrective therapies are allowed within the first 14 days of obtaining laboratory tests), as follows.

   ① Blood count: absolute neutrophil count (ANC) ≥ 1.5×109/L; platelet count (PLT) ≥ 75×109/L; hemoglobin level (HGB) ≥ 9.0 g/dL.

   ② Liver function: serum total bilirubin (TBIL) ≤2× upper limit of normal (ULN); alanine amino transferase (ALT) and aspartate aminotransferase (ST) ≤5×ULN; serum albumin ≥28 g/L; alkaline phosphatase (ALP) ≤5×ULN.

   (iii) Renal function: serum creatinine (Cr) ≤ 1.5×ULN or creatinine clearance (CCr) ≥ 50 mL/min (Cockcroft-Gault formula); urine routine results show urine protein <2+; for patients with urine protein ≥2+ at baseline, 24-hour urine collection and 24-hour urine protein quantification <1g should be performed.

   ④ Coagulation: International normalized ratio (INR) and activated partial thromboplastin time (APTT) ≤ 1.5 times ULN.
10. Female patients of childbearing age or male patients whose sexual partners are women of childbearing age are required to use effective contraception throughout the treatment period and for 6 months after the last dose.
11. Sign a written informed consent form and be able to comply with protocol visits and related procedures.

Exclusion Criteria:

1. Patients with hepatocellular carcinoma who have received prior treatment with carrilizumab or any other PD-L1 or PD-1 antagonist, or who have participated in a phase III study with apatinib after receiving systemic therapy.
2. Subjects with any active autoimmune disease or history of autoimmune disease, including but not limited to: hepatitis, pneumonia, uveitis, colitis (inflammatory bowel disease), pituitary inflammation, vasculitis, nephritis, hyperthyroidism and hypothyroidism, except vitiligo or resolved childhood asthma/atopic disease. Patients with asthma requiring intermittent use of bronchodilators or other medical interventions should also be excluded.
3. Subjects with systemic or absorbable topical corticosteroids requiring immunosuppressive drugs or immunosuppressive doses. Prednisone or equivalent doses greater than 10 mg/day are contraindicated for 2 weeks prior to dosing. Corticosteroids for intravenous contrast allergy prophylaxis are permitted.
4. Persons with known or suspected allergic reactions to any component of the Karelixu formulation.
5. Central nervous system (CNS) metastases with clinical signs (including cerebral edema, steroid requirements, or progressive disease). Subjects receiving treatment for brain or meningeal metastases must be clinically stable (no evidence of new or enlarged metastases on magnetic resonance imaging [MRI] at least 4 weeks apart) and have discontinued treatment with systemic steroid immunosuppressive doses (>10 mg/day of prednisone or equivalent) at least 2 weeks prior to study drug.
6. Other malignancies (except cured basal cell carcinoma of the skin and cervical cancer)
7. Clinically significant cardiovascular disease, including but not limited to: severe acute myocardial infarction, unstable or severe angina, coronary artery bypass surgery, congestive heart failure (New York Heart Association (NYHA) class >2), ventricular arrhythmia requiring medical intervention, and left ventricular ejection fraction (LVEF) <50% within 6 months prior to enrollment.
8. Poorly controlled hypertension within 3 months: systolic blood pressure >140 mmHg, diastolic blood pressure >90 mmHg.
9. Subjects with bleeding tendency or on thrombolytic or anticoagulant therapy.
10. Subjects who have received systemic chemotherapy, radiotherapy, immunotherapy, hormonal therapy, surgery, or targeted therapy within 4 weeks (or equivalent to 5 half-lives, whichever is greater) prior to dosing or have any unresolved adverse event > Common Terminology Criteria for Adverse Events (CTCAE) Level 1 (allowing for unresolved stable chronic toxicity).
11. Subjects with clinically symptomatic ascites or pleural effusion that remains uncontrolled by therapeutic puncture and drainage.
12. History of gastrointestinal bleeding within 3 months or significant tendency to gastrointestinal bleeding such as: esophageal varices, locally active ulcerative lesions, gastric and duodenal ulcers, ulcerative colitis or gastrointestinal diseases such as portal hypertension or tumor resection with risk of bleeding
13. Severe bleeding (bleeding >30 ml within 3 months), hemoptysis (>5 ml within 4 weeks) or thromboembolic events (within 12 months, including stroke events and/or transient ischemic attacks).
14. Active infection or fever of unknown origin >38.5°C during the screening visit or on the first scheduled dosing date (patients with fever due to tumor may be included at the discretion of the investigator)
15. History of pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, radiation pneumonia, drug-related pneumonia, or severely impaired lung function.
16. History of immunodeficiency including human immunodeficiency virus (HIV) positive, or other acquired or congenital immunodeficiency disease, or active hepatitis (transaminases not meeting inclusion criteria, hepatitis B virus (HBV) DNA ≥ 104/ml or hepatitis C virus (HCV) RNA ≥ 103/ml (or higher). Chronic hepatitis B virus carriers with HBV DNA <2000 IU/ml (<104/ml) must receive antiviral therapy throughout the study.
17. Subjects who have participated in other clinical trials or completed other clinical trials within 4 weeks.
18. Subjects who may be receiving other anti-tumor systemic therapy during the study.
19. Subjects who may have received a vaccine during the study period or who have previously received a vaccine within 4 weeks.
20. History of psychiatric disorder or psychotropic substance abuse.
21. Any other medical, psychiatric or social condition that, in the opinion of the investigator, may affect the subject's rights, safety, welfare or ability to sign informed consent, cooperate and participate in the study or interfere with the interpretation of the results.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-10-31 (Estimated)

PRIMARY OUTCOMES:
objective response rate(ORR) | 1 year
  The proportion of patients with tumor volume reduction up to a pre-specified value and able to maintain the minimum time requirement is the sum of the proportion in complete and partial remission
disease control rate(DCR) | 1 year
  The number of cases with remission and stable lesions after treatment as a percentage of evaluable cases that were maintained for at least 4 weeks.
overall survival(OS) | 1 year
  The time interval from the start of treatment until the patient's death (from any cause)
progression-free survival(PFS) | 1 year
  Time interval from the start of treatment until disease progression (including death)
Number of participants with treatment-related adverse events as assessed by NCI-CTCAE 5.0." | 1 year
  Side effects due to immunotherapy

SECONDARY OUTCOMES:
Change in tumor volume before and after treatment | 24 weeks
  The efficacy of the study will be evaluated based on the imaging results and evaluation criteria for efficacy of solid tumorssolid tumors (RECISTv1.1).

CONTACTS AND LOCATIONS:
Overall Officials: Chan Xie, PhD, Principal Investigator — Third Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- The Third Affiliated Hospital of Sun Yat-Sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Meng X, Liu X, Guo X, Jiang S, Chen T, Hu Z, Liu H, Bai Y, Xue M, Hu R, Sun SC, Liu X, Zhou P, Huang X, Wei L, Yang W, Xu C. FBXO38 mediates PD-1 ubiquitination and regulates anti-tumour immunity of T cells. Nature. 2018 Dec;564(7734):130-135. doi: 10.1038/s41586-018-0756-0. Epub 2018 Nov 28. PMID 30487606
- [Background] Ruiz de Galarreta M, Bresnahan E, Molina-Sanchez P, Lindblad KE, Maier B, Sia D, Puigvehi M, Miguela V, Casanova-Acebes M, Dhainaut M, Villacorta-Martin C, Singhi AD, Moghe A, von Felden J, Tal Grinspan L, Wang S, Kamphorst AO, Monga SP, Brown BD, Villanueva A, Llovet JM, Merad M, Lujambio A. beta-Catenin Activation Promotes Immune Escape and Resistance to Anti-PD-1 Therapy in Hepatocellular Carcinoma. Cancer Discov. 2019 Aug;9(8):1124-1141. doi: 10.1158/2159-8290.CD-19-0074. Epub 2019 Jun 11. PMID 31186238
- [Background] Chemnitz JM, Parry RV, Nichols KE, June CH, Riley JL. SHP-1 and SHP-2 associate with immunoreceptor tyrosine-based switch motif of programmed death 1 upon primary human T cell stimulation, but only receptor ligation prevents T cell activation. J Immunol. 2004 Jul 15;173(2):945-54. doi: 10.4049/jimmunol.173.2.945. PMID 15240681
- [Background] Riley JL. PD-1 signaling in primary T cells. Immunol Rev. 2009 May;229(1):114-25. doi: 10.1111/j.1600-065X.2009.00767.x. PMID 19426218
- [Background] Janney A, Powrie F, Mann EH. Host-microbiota maladaptation in colorectal cancer. Nature. 2020 Sep;585(7826):509-517. doi: 10.1038/s41586-020-2729-3. Epub 2020 Sep 23. PMID 32968260
- [Background] Ma C, Han M, Heinrich B, Fu Q, Zhang Q, Sandhu M, Agdashian D, Terabe M, Berzofsky JA, Fako V, Ritz T, Longerich T, Theriot CM, McCulloch JA, Roy S, Yuan W, Thovarai V, Sen SK, Ruchirawat M, Korangy F, Wang XW, Trinchieri G, Greten TF. Gut microbiome-mediated bile acid metabolism regulates liver cancer via NKT cells. Science. 2018 May 25;360(6391):eaan5931. doi: 10.1126/science.aan5931. PMID 29798856
- [Background] Routy B, Le Chatelier E, Derosa L, Duong CPM, Alou MT, Daillere R, Fluckiger A, Messaoudene M, Rauber C, Roberti MP, Fidelle M, Flament C, Poirier-Colame V, Opolon P, Klein C, Iribarren K, Mondragon L, Jacquelot N, Qu B, Ferrere G, Clemenson C, Mezquita L, Masip JR, Naltet C, Brosseau S, Kaderbhai C, Richard C, Rizvi H, Levenez F, Galleron N, Quinquis B, Pons N, Ryffel B, Minard-Colin V, Gonin P, Soria JC, Deutsch E, Loriot Y, Ghiringhelli F, Zalcman G, Goldwasser F, Escudier B, Hellmann MD, Eggermont A, Raoult D, Albiges L, Kroemer G, Zitvogel L. Gut microbiome influences efficacy of PD-1-based immunotherapy against epithelial tumors. Science. 2018 Jan 5;359(6371):91-97. doi: 10.1126/science.aan3706. Epub 2017 Nov 2. PMID 29097494
- [Background] Gopalakrishnan V, Spencer CN, Nezi L, Reuben A, Andrews MC, Karpinets TV, Prieto PA, Vicente D, Hoffman K, Wei SC, Cogdill AP, Zhao L, Hudgens CW, Hutchinson DS, Manzo T, Petaccia de Macedo M, Cotechini T, Kumar T, Chen WS, Reddy SM, Szczepaniak Sloane R, Galloway-Pena J, Jiang H, Chen PL, Shpall EJ, Rezvani K, Alousi AM, Chemaly RF, Shelburne S, Vence LM, Okhuysen PC, Jensen VB, Swennes AG, McAllister F, Marcelo Riquelme Sanchez E, Zhang Y, Le Chatelier E, Zitvogel L, Pons N, Austin-Breneman JL, Haydu LE, Burton EM, Gardner JM, Sirmans E, Hu J, Lazar AJ, Tsujikawa T, Diab A, Tawbi H, Glitza IC, Hwu WJ, Patel SP, Woodman SE, Amaria RN, Davies MA, Gershenwald JE, Hwu P, Lee JE, Zhang J, Coussens LM, Cooper ZA, Futreal PA, Daniel CR, Ajami NJ, Petrosino JF, Tetzlaff MT, Sharma P, Allison JP, Jenq RR, Wargo JA. Gut microbiome modulates response to anti-PD-1 immunotherapy in melanoma patients. Science. 2018 Jan 5;359(6371):97-103. doi: 10.1126/science.aan4236. Epub 2017 Nov 2. PMID 29097493
- [Background] Matson V, Fessler J, Bao R, Chongsuwat T, Zha Y, Alegre ML, Luke JJ, Gajewski TF. The commensal microbiome is associated with anti-PD-1 efficacy in metastatic melanoma patients. Science. 2018 Jan 5;359(6371):104-108. doi: 10.1126/science.aao3290. PMID 29302014
- [Background] Mager LF, Burkhard R, Pett N, Cooke NCA, Brown K, Ramay H, Paik S, Stagg J, Groves RA, Gallo M, Lewis IA, Geuking MB, McCoy KD. Microbiome-derived inosine modulates response to checkpoint inhibitor immunotherapy. Science. 2020 Sep 18;369(6510):1481-1489. doi: 10.1126/science.abc3421. Epub 2020 Aug 13. PMID 32792462
- [Background] Zheng Y, Wang T, Tu X, Huang Y, Zhang H, Tan D, Jiang W, Cai S, Zhao P, Song R, Li P, Qin N, Fang W. Gut microbiome affects the response to anti-PD-1 immunotherapy in patients with hepatocellular carcinoma. J Immunother Cancer. 2019 Jul 23;7(1):193. doi: 10.1186/s40425-019-0650-9. PMID 31337439
- [Background] Jiang Y, Han QJ, Zhang J. Hepatocellular carcinoma: Mechanisms of progression and immunotherapy. World J Gastroenterol. 2019 Jul 7;25(25):3151-3167. doi: 10.3748/wjg.v25.i25.3151. PMID 31333308
- [Background] Schwabe RF, Greten TF. Gut microbiome in HCC - Mechanisms, diagnosis and therapy. J Hepatol. 2020 Feb;72(2):230-238. doi: 10.1016/j.jhep.2019.08.016. PMID 31954488